CLINICAL TRIAL: NCT04628208
Title: Assess the Performance of Spartan COVID-19 V2 System in a Clinical Setting in Comparison to a Laboratory (Standard of Care (SOC)) PCR Method (Canada Alternate)
Brief Title: Clinical Study Spartan COVID-19 V2 System (Canada Alternate)
Status: Completed | Type: Observational
Sponsor: Spartan Bioscience Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VNV-00635
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative for COVID-19: Subject determined to be negative for COVID-19 by the standard of care nasopharyngeal swab-based SARS-CoV-2 RT-PCR test.
  Interventions: Diagnostic Test: Spartan COVID-19 v2 System
- Positive for COVID-19: Subject determined to be positive for COVID-19 by the standard of care nasopharyngeal swab-based SARS-CoV-2 RT-PCR test.
  Interventions: Diagnostic Test: Spartan COVID-19 v2 System

INTERVENTIONS:
Diagnostic Test: Spartan COVID-19 v2 System — A nasopharyngeal swab sample analyzed on the Spartan COVID-19 v2 System for the detection of SARS-CoV-2.

SUMMARY:
This multicentre prospective study will enroll a sufficient number of patients to afford approximately 30 positives and > 30 negatives (as determined by the SOC - Comparator method) in the United States and/or Canada. One to three sites in the Canada will participate over an approximate 6-week enrolment period. The actual enrolment period will be dependent upon prevalence of Covid-19, and site set up. Once positives sample size is achieved, expected SARC-CoV-2 negative subjects will be permitted.

Once subjects are consented and recruited for the study, up to three (3) study-specific nasopharyngeal samples for each patient will be collected by trained operators at the clinical site: a single SOC swab, and two (2) Spartan swabs where the second swab is optional and used when the first Spartan swab test does not produce a positive or negative result ("inconclusive").

The first swab sample will be tested at the clinical site according to standard of care protocols currently in place for the sites' nasopharyngeal swab-based SARS-CoV-2 RT-PCR testing. The second nasopharyngeal sample will be tested at the site using the Spartan COVID-19 v2 System. A third, optional nasopharyngeal sample, if collected, will be tested using the Spartan COVID-19 v2 System only when the test conducted with the second nasopharyngeal swab does not produce a positive or negative result.

ELIGIBILITY:
Inclusion Criteria:

* Suspected SARS-CoV-2 infection by a healthcare provider, and whose first symptoms presented ≤ 7 days of onset; or
* Suspected SARS-CoV-2 infection from the same household of a person who tested positive for SARS-CoV-2 using an authorized test; or
* Known positive SARS-CoV-2 infection using an authorized test, and whose first symptoms presented ≤ 7 days of onset; or
* Expected negative SARS-CoV-2 infection - individuals with no symptoms or a recent negative result by an authorized test.

Exclusion Criteria:

* Vulnerable populations (e.g., women with pregnancy, institutionalized individual) as deemed inappropriate for study by the site investigator
* Individuals with self-reported nosebleed within 24 hours of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to clinical study sites with symptoms of SARS-CoV-2 or suspected of SARS-Cov-2 infection by a healthcare provider
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Percent Agreement between SOC test and Spartan COVID-19 test | 24 hours
  Overall percent agreement between the test results generated by the Spartan COVID-19 v2 System and the nasopharyngeal swab-based SARS-Cov-2 test currently in use at the clinical site (SOC test)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa hospital, Ottawa, Ontario, Canada